CLINICAL TRIAL: NCT06104501
Title: Validation of the Blood Pressure Monitoring Function of a Fingertip Photoplethysmography
Brief Title: Validation of the Blood Pressure Monitoring Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RadiRad Co., Ltd. (Industry)
Collaborators: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Validation of Blood Pressure
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Blood Pressure
Keywords: Artificial Intelligence(AI) Algorithm; blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RadiHeart — The participants' blood pressure will be measured multiple times by both the mercury sphygmomanometer and RadiHeart, by using the same arm sequential method.

SUMMARY:
High blood pressure is a major risk factor for cardiovascular diseases, stroke, and kidney disorders. Accurate blood pressure monitoring is crucial for the diagnosis, treatment, and prevention of complications related to high blood pressure. In recent years, due to the rapid development of wearable devices and mobile technology, wearable blood pressure monitors have gradually become a non-invasive and convenient method for blood pressure monitoring. However, the accuracy of these devices has not been fully established. This study aims to validate the performance of RadiHeart (an application program) in blood pressure measurement.

DETAILED DESCRIPTION:
Following the ISO 81060-2:2018 standard, the accuracy of RadiHeart will be evaluated by comparing the blood pressure values obtained by the device with those measured by a conventional mercury sphygmomanometer. This research is expected to recruit 170 adults aged 20 and above. All participants will undergo blood pressure measurements using both RadiHeart and a mercury sphygmomanometer. Participants will operate RadiHeart under the guidance of the testing personnel, while the mercury sphygmomanometer will be operated by trained healthcare professionals. The blood pressure measurement results from both devices will be recorded simultaneously, and the consistency between the blood pressure values measured by RadiHeart and the traditional mercury sphygmomanometer will be compared to validate the accuracy of the blood pressure application.

ELIGIBILITY:
Inclusion Criteria:

The subjects should be aged 20 or older, with an equal gender distribution of 50% male and 50% female. From this group, 85 subjects with reasonable data values will be selected, with a requirement that at least 30% of them are male and at least 30% are female. Additionally, they must meet the following blood pressure conditions:

1. At least 5% (5 individuals) of the participants should have reference systolic blood pressure readings ≥ 160 mmHg (21.33 kPa).
2. At least 20% (17 individuals) of the participants should have reference systolic blood pressure readings ≥ 140 mmHg (18.66 kPa).
3. At least 5% (5 individuals) of the participants should have reference systolic blood pressure readings ≤ 100 mmHg (13.33 kPa).
4. At least 5% (5 individuals) of the participants should have reference diastolic blood pressure readings ≤ 60 mmHg (8.0 kPa).
5. At least 20% (17 individuals) of the participants should have reference diastolic blood pressure readings ≥ 85 mmHg (11.33 kPa).
6. At least 5% (5 individuals) of the participants should have reference diastolic blood pressure readings ≥ 100 mmHg (13.33 kPa).

Exclusion Criteria:

1. Pregnant.
2. Having any of the following conditions:

   * Arrhythmia
   * Medical assessment indicates that poor blood circulation would affect the blood pressure data collection.
   * Involuntary hand movements that would affect the blood pressure data collector.
   * Nail polish on the light sensor area of the fingertip oximeter.
   * Other conditions as determined by a physician that make the individual unsuitable for participation in the trial.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This trial expects to enroll 170 participants. The subjects should be aged 20 or older, with an equal gender distribution of 50% male and 50% female. From this group, 85 subjects with reasonable data values will be selected, with a requirement that at least 30% of them are male and at least 30% are female.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in blood pressure (mean) | 1 hour per individual
  The mean value of the differences in blood pressure measured by RadiHeart and the reference sphygmomanometer should be within or equal to ±5.0 mmHg.
Difference in blood pressure (standard deviation) | 1 hour per individual
  The standard deviation of the differences in blood pressure measured by RadiHeart and the reference sphygmomanometer should be no greater than 8.0 mmHg.

IPD SHARING:
Plan to Share IPD: No